CLINICAL TRIAL: NCT01088087
Title: Effect of Colostrum Administration on Improving Gut Permeability and Serum Endotoxin Level in Chronic Alcohol Drinkers With Hepatic Dysfunction
Brief Title: Effect of Colostrum on Gut Permeability and Endotoxin Level in Chronic Alcoholic Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Cell Biotech Co., Ltd. (Industry)
Responsible Party: Yonsei University, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GangnamSH
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2009-11

CONDITIONS: Leaky Gut Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colostrum (Placebo Comparator)
  Interventions: Dietary Supplement: colostrum
- Sugar pill (No Intervention)

INTERVENTIONS:
Dietary Supplement: colostrum — colostrum, 2g, 2 times a day, for 3 weeks
  Other Names: Mucoba
  Arms: Colostrum

SUMMARY:
Chronic alcohol ingestion is related with leaky gut syndrome. Colostrum is well-studied that it has a effect of decreasing the degree of leaky gut syndrome.

So the investigators are planning to find out whether Colostrum has a effect of decreasing the degree of leaky gut syndrome.

DETAILED DESCRIPTION:
We randomly sort the participant as placebo group and colostrum group. Each group consists of 17 people. and the duration of our study for one participant is 3 weeks. (Participant takes colostrum for 3 weeks.)

When a person gets leaky gut syndrome, his or her endotoxin and lactulose/mannitol ratio (L/M ratio, in urine) can elevate.

So We will compare the value of those two parameters and LFT. etc. after the administration of colostrum or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men aged over 20 who's alcohol consumption per day is 20.0gram average

  * He must agree to participate this trial voluntarily.
* Liver function test within 3 months :

AST more than 30 or ALT more than 33 or Gamma-GT more than 46

* Men who have result of Ultra-sono result of abdomen without Liver cirrhosis

Exclusion Criteria:

* Hepatitis B or C , liver cirrhosis patient
* Men who have undergo bowel operation
* Men who are taking NSAIDs
* Periodontitis or GERD or other G-I tract infection within 2 weeks before enrollment
* Men who have been given anticancer drug within one year
* Men who have been given antibiotics within 2 weeks
* Creatinine level >= 1.4mg/dl
* Men who are taking G-I motility drugs or anti-ulcer drug
* Milk allergy

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
endotoxin | 1st visit and 3 weeks after 1st visit

SECONDARY OUTCOMES:
lactulose/mannitol ratio | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Shim, Master, Study Director — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital : Family medicine department, Seoul, South Korea